CLINICAL TRIAL: NCT04973982
Title: ENvarsus for Impaired Glucose Tolerance Post REnal transplAnT
Acronym: ENTREAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of capacity
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012280
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-07

CONDITIONS: Renal Transplant Failure
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single centre, randomised parallel-group controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENVARSUS (Active Comparator): ENVARSUS used as per licence
  Interventions: Drug: Envarsus
- ADOPORT (Active Comparator): ADOPTION used as per licence
  Interventions: Drug: Adoport

INTERVENTIONS:
Drug: Envarsus — 3 month treatment, given once daily, oral tablet. Dose titrated according to levels target 6-10ng/ml
  Arms: ENVARSUS
Drug: Adoport — 3 month treatment, given twice daily, oral tablet. Dose titrated according to levels target 6-10ng/ml
  Other Names: Tacrolimus
  Arms: ADOPORT

SUMMARY:
Our hypothesis is that switching from the current standard of care twice daily Adoport (Tacrolimus) to once daily Envarsus (tacrolimus) in patients who have impaired glucose tolerance post-transplant will lead to an improvement in their glucose tolerance, and may reduce the subsequent incidence of PTDM.

DETAILED DESCRIPTION:
Kidney transplantation is widely held to be the optimal form of renal replacement therapy for patients with end-stage renal disease, leading to a longer survival and improved quality of life in patients receiving a renal transplant compared to those that remain on dialysis. However renal transplantation brings with it a new set of challenges for the clinician. One of the most important of these is post-transplant diabetes mellitus (PTDM). The prevalence of PTDM has increased over time and may occur in up to a third of all post-transplant patients making it a critical challenge for transplant physicians.

PTDM represents a significant risk factor to both patient and graft survival, with some studies suggesting an increase of 60% in graft failure and an almost 90% increase in mortality. This morbidity and mortality is due to the greatly increased risk of cardiovascular disease associated with PTDM. In addition to the clinical consequences of PTDM for patients, there is also a huge economic impact on healthcare, with a diagnosis of PTDM doubling the cost of healthcare for a transplant patient.

Important risks factors for PTDM include: Black/Asian race, male sex, older patients, receipt of a 'Donation after cardiac death' kidney, family history of diabetes, BP, raised body-mass index, Hepatitis C disease, Cytomegalovirus (CMV) viraemia, hyperparathyroidism, low HDL cholesterol, and hypomagnesaemia.

In addition, PTDM is caused by multiple factors associated with renal transplantation. Steroid use impairs pancreatic beta-cell function, induces gluconeogenesis and glycolysis, inhibits glycogenesis and leads to insulin resistance. Tacrolimus, a calcineurin inhibitor (CNI), has been associated with increased rates of PTDM when compared to other CNIs (i.e. cyclosporine). It leads to hyperglycaemia via reduction of pancreatic insulin secretion and a reduction of GLUT-4 mediated glucose uptake into cells. In addition, it may directly cause beta cell toxicity and down regulate insulin gene expression. High tacrolimus concentrations have been associated with the development of PTDM; however, due to its enhanced efficacy in prevention of acute and chronic rejection, it has become the most widely used immunosuppressive medication in renal transplantation.

Over 30% of patients post renal transplant have evidence of impaired glucose tolerance (IGT). IGT is a key step in the development of PTDM and an opportunity for intervention to prevent the development of PTDM.

Higher peak tacrolimus levels have been associated with islet cell damage leading to hyperglycaemia, with evidence that this damage may be reversible with changing tacrolimus exposure .

Not all tacrolimus based regimens may have the same side effects. Envarsus is a newer tacrolimus formulation, which has significantly altered pharmacokinetic properties and bioavailability compared to other tacrolimus based regimens.

Envarsus has significantly lower peak to trough ratios and a 30% lower peak concentration. Both of these unique properties may reduce the beta cell toxicity seen with older tacrolimus based regimens and lead to an improvement in impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria

1. Females or males aged 18 years and above
2. Having undergone renal transplantation within the previous 2 years
3. Current treatment with tacrolimus
4. Evidence of impaired glucose tolerance (defined as a blood glucose level between 7.8-11.1 mmol/L after a two hour oral glucose tolerance test)
5. Provision of written, informed consent prior to any study specific procedures

Exclusion Criteria

1. Unable to consent
2. Planning on becoming pregnant/unwilling to use highly effective contraception during the 3-month treatment period or breastfeeding.
3. Clinically significant history of abnormal physical and/or mental health as judged by the investigator other than conditions related to chronic kidney disease
4. History of Type 1 or Type 2 diabetes mellitus; or on treatment with anti-diabetic medications
5. Prior therapy with Envarsus
6. Exposure to an investigational drug withing the preceding 3 months, or 5 half-lives whichever is greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who normalise their IGT (defined as a blood glucose level between <7.8mmol/l) after a two-hour oral glucose tolerance test at three months after randomisation. | 3 months
  The proportion of patients who normalise their IGT (defined as a blood glucose level between <7.8mmol/l) after a two-hour oral glucose tolerance test at three months after randomisation.

SECONDARY OUTCOMES:
Change in HOMA-IR test between 0 and 3 months post-randomisation This parameter will be compared on the ITT dataset using unpaired T test. P values of < 0.05 will be considered statistically significant | 3 month
  Change in HOMA-IR test between 0 and 3 months post-randomisation
Proportion of patients developing PTDM during the study | 3 month
  Proportion of patients developing PTDM during the study as defined by a positive two-hour OGTT >11.1 mmol/L at 3 months
Change in HbA1c between baseline and 3 months This parameter will be compared on the ITT dataset using unpaired T test. P values of < 0.05 will be considered statistically significant. | 3 month
  Change in HbA1c between baseline and 3 months
Change in eGFR between baseline and 3 months This parameter will be compared on the ITT dataset using unpaired T test. P values of < 0.05 will be considered statistically significant. | 3 month
  Change in eGFR between baseline and 3 months
Change in fasting blood sugar between randomisation and month 3 This parameter will be compared on the ITT dataset using unpaired T test. P values of < 0.05 will be considered statistically significant. | 3 month
  Change in fasting blood sugar between randomisation and month 3
Change in 2h OGTT blood result between randomisation and month 3 This parameter will be compared on the ITT dataset using unpaired T test. P values of < 0.05 will be considered statistically significant. | 3 month
  Change in 2h OGTT blood result between randomisation and month 3
Safety endpoints: SAEs, AEs AE and SAE will be categorised into categories as per CRF. | 3 month
  Frequency of SAEs and AEs occurring during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
aggregated data will be shared